CLINICAL TRIAL: NCT06260319
Title: Decoding Developmental Disorders in Humams, Devodecode
Brief Title: Decoding Developmental Disorders in Humams
Acronym: devodecode
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Imagine Institute (Other); Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Other Study IDs: C19-64
Record Dates: First submitted 2024-01-12; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Genetic Diseases
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole genome sequencing (WGS) and bioinformatics analysis Functional validation Genome-Epigenome-Phenome Associations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Whole genome sequencing and Genome-Epigenome-Phenome Associations — * Whole genome sequencing (WGS) and bioinformatics analysis
  * Functional validation
  * Genome-Epigenome-Phenome Associations

SUMMARY:
The DEVO-DECODE project aims to align our currently limited knowledge currently limited knowledge of the genetic architecture of developmental with our more advanced knowledge of their "phenome".

To this end, we aim to establish a homogeneous cohort of patients with with developmental disorders to identify new genetic variants genetic variants, and thus study the association between developmental and genetic variants. Secondary objectives are:2

* Carry out WGS studies not only to refine exosomal sequencing data exome sequencing data, but above all to identify and validate non-coding non-coding DNA alterations, in both transcribed and non-transcribed transcribed or non-transcribed genomic domains
* Develop precise preclinical models for functional studies of pathophysiological pathways

DETAILED DESCRIPTION:
Developmental disorders, which encompass congenital anomalies and intellectual disabilities - including autism spectrum disorders - constitute a vast group of pathologies, caused by a complex set of genetic and environmental factors. They can affect several organs or tissues, such as brain abnormalities, head and neck malformations, heart defects, skeletal disorders and ophthalmological or hearing pathologies. They occur in around 2-3% of live births - affecting around 150,000 newborns every year in Europe (1). These pathologies are associated with high morbidity and mortality rates. They were responsible for 632,000 deaths worldwide in 2013 (2), representing a major social, economic and health problem.

Together, these diseases represent a considerable challenge in terms of medical care and genetic counseling, underlining the major deficits in fundamental and clinical knowledge to date.

At the Hôpital Necker-Enfants malades and the Institut des Maladies Génétiques Imagine, between 20,000 and 25,000 patients suffering from a wide range of developmental disorders are treated every year. Multidisciplinary consultations, together with state-of-the-art genomic investigations such as comparative genome hybridization (CGH) and whole exome sequencing (WES), provide the research and clinical teams involved with in-depth knowledge of the natural history of these diseases and the phenotypes of affected patients, as well as a better understanding of their genetic basis. Despite this, the rate of unknown diagnoses is very high (over 65-70% of cases remain without a distinct pathophysiological label), due to both the heterogeneity of these diseases and the complexity of their genetic architecture, probably involving non-coding DNA in many cases. Studying this non-coding DNA therefore requires technologies such as whole genome sequencing (WGS).

The main aim of the DEVO-DECODE project is to align our currently limited knowledge of the genetic architecture of developmental disorders with our more advanced knowledge of their "phenome". To meet this challenge,we propose to draw on the expertise and resources available within the research and clinical teams at Institut Imagine and Hôpital Necker, in order to:

1. create well-characterized, homogeneous cohorts.
2. systematize the collection of samples from patient care for biobanking and other studies.
3. carry out WGS studies not only to refine exome sequencing data, but above all to identify and validate non-coding DNA alterations, in both transcribed and non-transcribed genomic domains.
4. develop precise preclinical models for functional studies of candidate pathophysiological pathways.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adult patients with hereditary diseases and relatives who have consented to the storage of their biological samples in the Institut Imagine's declared biological collections.
* Pediatric and adult patients with hereditary diseases and relatives who have been informed of the research project and who have not objected to the re-use of their data and biological samples samples

Exclusion Criteria:

-

Ages: 1 Year to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients with hereditary diseases and related who have consented to the storage of their biological samples biological samples as part of the Institut Imagine's declared biological
  Institut Imagine, selected on the basis of the following criteria :
  - negative preliminary CGH or WES sequencing data
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Primary objectives | up to 2 years
  Establish a homogeneous cohort of patients with developmental developmental disorders to identify new genetic variants, and thus study the association between developmental pathologies and genetic variants.

SECONDARY OUTCOMES:
secondary objectives 1 | up to 2 years
  Carry out WGS studies not only to refine exome sequencing data exome sequencing data, but above all to identify and validate non-coding non-coding DNA alterations, in both transcribed and non-transcribed transcribed or non-transcribed genomic domains
secondary objectives 2 | up to 2 years
  Develop precise preclinical models for functional studies of pathophysiological pathways.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Imagine, Paris, France